CLINICAL TRIAL: NCT03302689
Title: The Double-blind, Randomized Controlled Trial: Comparison of Levobupivacaine and Ropivacaine for Postoperative Analgesia TAP-block After Caesarean Section
Brief Title: Comparison Levobupivacaine and Ropivacaine for TAP-block After Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandr Ronenson (Other)
Responsible Party: Sponsor-Investigator, Alexandr Ronenson, Head of department of Anaesthesiology and Intensive Care Unit, Tver Regional Perinatal Center
Organization: Tver Regional Perinatal Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LeRoTAP
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Pain, Postoperative
Keywords: TAP-block; VAS of pain; Cesarean section; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two groups of women after cesarean section under spinal anesthesia
Who Masked: Participant, Investigator
Masking Description: Women after the operation do not know what drug they injected with TAP-block The researcher does not know what type of drug is injected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): TAP-block with Ropivacaine Solution
  Interventions: Drug: Ropivacaine Solution
- Levobupivacaine (Experimental): TAP-block with Levobupivacaine Solution
  Interventions: Drug: Levobupivacaine Solution

INTERVENTIONS:
Drug: Levobupivacaine Solution — TAP-block with Levobupivacaine 0,3% - 25 ml from each side
  Other Names: Levo
  Arms: Levobupivacaine
Drug: Ropivacaine Solution — TAP-block with Ropivacaine 0,3% - 25 ml from each side
  Other Names: Rop
  Arms: Ropivacaine

SUMMARY:
Randomized, double-blind, controlled trial: a comparison of Levobupivacaine and Ropivacaine for postoperative analgesia using TAP-block

Objectives:

1. VAS score during the first 12 hours
2. Determine which drug is more effective for postoperative analgesia in the first 12 hours after surgery
3. Side effects

DETAILED DESCRIPTION:
For TAP-block was used Hirokain® (Levobupivacaine) . Injectable solution 7.5 mg / ml; ampoule polypropylene 10 ml, a pack of cardboard 10; No. ЛП-003106, 2015-07-21 to 2020-07-21 from EbbVi Ltd. (Russia); manufacturer: Kurida AS (Norway); Packer: AbbVi S.r.l. (Italy), or Ropivacaine Kabi (Ropivacaine Kabi) (Ropivacaine) Solution for injection 7.5 mg / ml; ampoule polypropylene 1 10 ml, a pack of cardboard 5; EAN code: 4607085481524; No. ЛП-002897, 2015-03-04 to 2020-03-04 from Fresenius Kabi Deutschland GmbH (Germany); manufacturer: Fresenius Kabi Norge (Norway).

Both preparations were diluted to a volume of 50 ml, at a concentration of 3 mg / ml.

It was performed by TAP-block in-plain with a 22G needle Quincke, on both sides, and 25 ml on each side was injected.

The pain syndrome was assessed with admission, and every 2 hours during the first 12 hours after the operation, using a digital scale on the VAS.

All patients received NSAIDs (Ketorol 3 mg IV every 6 hours from admission)

Additionally:

Paracetamol IV infusion 100 ml with VAS = 4 score, lockout time 6 hours Tramadol 5% - 2 ml IM with VAS = or > 5 score, lockout time 6 hours

ELIGIBILITY:
Inclusion Criteria:

* Cesarean section pfannenstiel incision under spinal anesthesia
* Spinal anesthesia with Bupivacaine heavy 0,5%
* Without any adjuvants

Exclusion Criteria:

* Any other anesthesia exept spinal
* Any other surgical incision

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Level of pain | 12 hours
  Measurement of pain on a VAS scale (from 0 to 10 points)

SECONDARY OUTCOMES:
The need for additional analgesics (Paracetamol, Tramadol) | 12 hours
  Paracetamol IV infusion 100 ml with VAS = 4 score, Tramadol 5% - 2 ml IM with VAS = 5 scores

CONTACTS AND LOCATIONS:
Locations (1):
- Tver Regional Perinatal Center, Tver', Russia

IPD SHARING:
Plan to Share IPD: No